CLINICAL TRIAL: NCT01405443
Title: Simulator Training for Gastrointestinal Endoscopy - How Much Simulator Training is Required to Acquire Proficiency in Gastrointestinal Endoscopy?
Brief Title: Simulator Training for Gastrointestinal Endoscopy
Status: Terminated | Type: Observational
Why Stopped: invalid data
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Prof. Dr. Thomas Roesch, Universitätsklinikum Hamburg-Eppendorf, Endoscopy department, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: UKE Hamburg Endoscopy PV3656
Record Dates: First submitted 2011-04-15; First posted 2011-07-29 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Performance of Inappropriate Operation
Keywords: Simulator training; Flexible endoscopy; Gastrointestinal endoscopy; Colonoscopy; Training; Performance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Basic training: Theory lecture esophagogastroduodenoscopy (EGD). One hour simulator training for EGD. 30 minutes supervised training. Supervised endoscopy. Theory lecture Colonoscopy. One hour simulator training for Colonoscopy. 30 minutes supervised training. Supervised endoscopy. Group will be followed up for 2 weeks training time.
- Intermediate training: Theory lecture EGD. Three hours simulator training for EGD. 60 minutes supervised training. Supervised endoscopy. Theory lecture Colonoscopy. Three hours simulator training for Colonoscopy. 60 minutes supervised training. Supervised endoscopy. Group will be followed up for 4 weeks training time.
- Extended training: Theory lecture EGD. Five hours simulator training for EGD. 90 minutes supervised training. Supervised endoscopy. Theory lecture Colonoscopy. Five hours simulator training for Colonoscopy. 90 minutes supervised training. Supervised endoscopy. Group will be followed up for 6 weeks training time.

SUMMARY:
This is a randomized controlled trial evaluating three training intervals using an endoscopy simulator for novices and comparing performance after training.

DETAILED DESCRIPTION:
Randomized controlled trial evaluating different training intervals on an endoscopy simulator and comparing performance using a validated score (Global assessment of Gastrointestinal Endoscopic Skills). Physicians participating in the study are novices with no previous experience in flexible endoscopy. Subjects are randomized into three different training arms. Proficiency scores will be evaluated by a supervising physician blinded to group allocation.

ELIGIBILITY:
Physicians in residency or fellowship programs requiring training in flexible endoscopy (gastroenterology, internal medicine, surgery) with no experience in flexible endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians in residency or fellowship programs requiring training in flexible endoscopy (gastroenterology, internal medicine, surgery) with no experience in flexible endoscopy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Validated proficiency score (GAGES "Global assessment for Gastrointestinal Endoscopy") for group one | Score is evaluated after one week training
  Score is a validated measuring tool based on intubation, scope navigation, ability to keep a clear endoscopic visualization and instrumentation.
Validated proficiency score (GAGES "Global assessment for Gastrointestinal Endoscopy") for group three | Score is evaluated after three weeks of training
  Score is a validated measuring tool based on intubation, scope navigation, ability to keep a clear endoscopic visualization and instrumentation.
Validated proficiency score (GAGES "Global assessment for Gastrointestinal Endoscopy") for group two | Score is evaluated after two weeks of training
  Score is a validated measuring tool based on intubation, scope navigation, ability to keep a clear endoscopic visualization and instrumentation.

SECONDARY OUTCOMES:
Simulator score | Score is evaluated after the training period (at one week for group 1, at 2 weeks for group 2, and at three weeks for group 3)
  Scores as evaluated by the Simbionix simulator software

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Sabrie N, Khan R, Plahouras J, Johnston BC, Scaffidi MA, Grover SC, Walsh CM. Virtual reality simulation training for health professions trainees in gastrointestinal endoscopy. Cochrane Database Syst Rev. 2025 Sep 8;9(9):CD008237. doi: 10.1002/14651858.CD008237.pub4. PMID 40919710